CLINICAL TRIAL: NCT01112566
Title: EASE MITRAL Expertise-based Assessment Study on Clinical Efficacy of Profile 3D in MITRAL Valve Annuloplasty
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Other Study IDs: BRC-CS-2010-03
Record Dates: First submitted 2010-04-27; First posted 2010-04-28 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Mitral Valve Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of the study is to identify the patients suffering from a mitral valve condition who benefit from the implantation of a Profile 3D annuloplasty ring in terms of acute and long-term relief of mitral valve regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* Indicated for a surgical repair for moderate to severe mitral valve regurgitation at rest (level 2 or higher);
* Willing to return to the hospital where the implantation originally occurred as part of the standard practice of care

Exclusion Criteria:

* Heavily calcified valves
* Valvular retraction with severely reduced mobility
* Active bacterial endocarditis
* Already participating in another investigational device study, possibly leading to bias and jeopardizing the scientific appropriate assessment of the study endpoints;
* Life expectancy of less than one year;
* Pregnant or desire to be pregnant within 12 months of the study treatment;
* Under 18 years or over 85 years of age.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population includes all patients suffering from mitral valve disease, indicated for a mitral valve repair procedure, either as a stand-alone procedure or concomitant to a coronary artery bypass grafting, an aortic replacement or tricuspid valve repair and/or the treatment of atrial fibrillation, and for which the surgeon considers the implantation of a Profile 3D annuloplasty product most appropriate to reconstruct the regurgitant valve.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2013-02; Primary Completion 2017-04-26 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Identify the patient population for which a Profile 3D Annuloplasty Ring is chosen to repair the mitral valve insufficiency. | screening
Assess the percentage of patients that are chronically relieved from mitral valve dysfunction | 6-12 months follow up
Determine the level of mitral valve regurgitation in patients | 6-12 months post-surgery

CONTACTS AND LOCATIONS:
Locations (7):
- London Health Sciences Centre, University Hospital, London, Ontario, Canada
- Nemocnice Ceske Budejovice A.S., České Budějovice, Czechia
- France (2):
  - Hôpital Haut - Leveque - CHU Pessac Cedex Bordeaux, Bordeaux
  - CHU de Nantes - Hôpital Nord Laennec, Nantes
- Germany (2):
  - Deutsches Herzzentrum München, München
  - SANA Herzchirurgie Stuttgart GmbH, Stuttgart
- Azienda Ospedaliero Universitaria Careggi, Florence, Italy

REFERENCES:
- [Derived] Doll N, Sheytanov V, Labrousse L, Chu MWA, Stefano P, Mokracek A, Baron O, Li S, Gunzinger R. Clinical performance of a three-dimensional saddle-shaped, rigid ring for mitral valve repair. Eur J Cardiothorac Surg. 2019 Feb 1;55(2):217-223. doi: 10.1093/ejcts/ezy215. PMID 29931248
- See also: Related Info — http://www.medtronic.com